CLINICAL TRIAL: NCT02250183
Title: A Comparison of Medihoney® Gel With Active Leptospermum Honey and Santyl® in the Treatment of Partial Thickness Burns
Brief Title: Medihoney and Santyl for Burn Injuries
Acronym: MSBI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was too slow due to strict inclusion criteria.
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: Integra LifeSciences Corporation (Industry); West Virginia University (Other)
Responsible Party: Principal Investigator, Christina Duncan, Professor of Psychology, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-021
Record Dates: First submitted 2014-09-15; First posted 2014-09-26 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Burns
Keywords: Medihoney; Santyl; Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Medihoney & Santyl (Other): Each patient will receive both interventions simultaneously, but on non-contiguous parts of the body that each consist of partial thickness burn injuries of similar depth. For example, if a patient presents with bilateral second-degree burns to the lower extremities, one leg will be treated with MEDIHONEY® GEL with Active leptospermum honey dressing, while the other leg will be treated with SANTYL® ointment dressing. MEDIHONEY® is the target treatment for this study, while SANTYL® is standard care.
  Interventions: Device: MEDIHONEY® GEL WITH ACTIVE LEPTOSPERMUM HONEY; Device: Santyl

INTERVENTIONS:
Device: MEDIHONEY® GEL WITH ACTIVE LEPTOSPERMUM HONEY — MEDIHONEY® GEL WITH ACTIVE LEPTOSPERMUM HONEY dressing is manufactured by the company Derma Sciences, Inc. and is a moist dressing made of Active Leptospermum Honey (+15) in combination with natural gelling agents. The gelling agents act to maintain the physical integrity and viscosity of the dressing, even in the presence of body heat and fluids. As a percentage of the overall dressing, MEDIHONEY® GEL dressings contains 80% honey. The dressing has a low pH and can help to lower the overall pH of wounds. The dressing also possesses a high osmotic potential, which assists in debridement.
  Other Names: Medihoney
Device: Santyl — SANTYL® Ointment is an FDA-approved sterile enzymatic debriding ointment which contains 250 collagenase units per gram of white petrolatum USP. The enzyme SANTYL® is derived from the fermentation by Clostridium histolyticum. It possesses the unique ability to digest collagen in necrotic tissue. SANTYL® Ointment is indicated for debriding chronic dermal ulcers and severely burned areas.

SUMMARY:
This study is designed to assess the efficacy of MEDIHONEY® Gel with Active leptospermum honey dressing relative to SANTYL® ointment dressing on time to heal, bacterial growth in the wound, patient satisfaction, and treatment costs in patients with partial thickness burns. The study has four hypotheses:

1. It is hypothesized that MEDIHONEY® Gel with Active leptospermum honey will result in significantly faster wound healing (i.e., fewer days) when compared to SANTYL®.
2. It is hypothesized that MEDIHONEY® Gel with Active leptospermum honey sites will yield significantly fewer positive cultures for Pseudomonas aeruginosa and other bacteria when compared to SANTYL® sites.
3. It is hypothesized that patients will provide significantly higher patient care satisfaction ratings regarding their MEDIHONEY® Gel with Active leptospermum honey sites when compared to ratings with regard to their SANTYL® sites.
4. It is hypothesized that treatment costs, across participants, will be significantly lower for MEDIHONEY® Gel with Active leptospermum honey than for SANTYL®.

DETAILED DESCRIPTION:
Researchers have examined the usefulness of honey as a treatment for a variety of wounds. Molan outlines some of the benefits of honey in the treatment of wounds, such as its effective antibacterial activity, debriding action, anti-inflammatory component, and antioxidant activity. In addition, the acidity of honey may improve wound healing by decreasing the pH of the wound and providing more oxygen, which ultimately helps to regenerate tissue .

Many studies have demonstrated the effectiveness of honey's antibacterial properties. For example, the antibacterial activity of honey has been shown to protect against multi-resistant strains of bacteria including multi-resistant staphylococcus aureus (MRSA) and Pseudomonas aeruginosa. In fact, research suggests that honey may be an effective antibacterial agent for bacteria that were resistant to up to 13 different antibiotics. Related specifically to burn injuries, results from another study indicated that honey may be an effective antibacterial agent and treatment option for burn injuries infected with or at risk for infection with Pseudomonas aeruginosa. Furthermore, unlike other antibiotics used in clinical care, the possibility of developing honey-resistant wound pathogens is rare, even when using high concentrations of honey, according to one study. Results from these studies provide strong evidence for the usefulness of honey's antibacterial activity in the treatment of wounds, including burn injuries.

In addition to its antibacterial properties, honey has been found to promote wound healing in patients with burn injuries. For example, one study compared the effectiveness of a honey dressing to silver sulfadiazene (SSD) on wound healing in 78 child and adult burn patients with first and second degree burns. According to the results from this study, patients treated with honey dressings had a significantly lower average duration of healing (in days) compared to patients treated with SSD. In addition, approximately half of the wounds treated with honey dressings became sterile within seven days while none of the wounds became sterile during this span of time for the patients who were treated with SSD. The authors of this study also reported that 30 of the 37 patients (81%) treated with honey achieved complete recovery (i.e., complete healing two months post-burn injury without scarring or contractures) compared to 15 out of 41 patients (37%) treated with SSD. Another study by Baghel and colleagues using a similar sample found comparable results. In this second study, patients who were treated with honey dressings were found to heal significantly faster, have sterile wounds in less time, and have better overall recoveries (i.e., fewer hypertrophic scars and contractures) when compared to those patients who were treated with SSD.

Another study compared honey and SSD on burn wound healing (i.e., improvement in burn wound size and re-epithelialization) in patients with superficial partial thickness burns. Patients included in this study had similar burns (e.g., second degree burns of similar depth) on comparable burned surface areas (e.g., right hand and left hand). In addition, patients in this study received both treatment options; that is, a patient's right hand was treated with honey while his/her left hand was treated with SSD. Results from this study indicated that the average healing time was significantly shorter for the body surfaces treated with honey. Interestingly, the wounds treated with honey were found to heal approximately two days faster than the wounds treated with SSD. Additionally, cultures of the wounds found that only six patients tested positive for Pseudomonas aeruginosa in the sites that were treated with honey compared to 27 patients in the sites treated with SSD. Two additional patients tested positive for Escherichia coli infection in the wound sites that were treated with SSD. The authors of this study concluded that honey was a more effective treatment for superficial partial thickness burns than SSD.

Taken together, these studies provide preliminary evidence that honey may be an effective treatment option for partial thickness burns, with benefits such as faster wound healing and wound sterilization. In addition, MEDIHONEY® is cleared by the FDA to maintain a moist environment conducive to wound healing. However, studies have yet to explore the generalizability of these findings to samples of patients with burn injuries in the United States, as all the previously cited studies were conducted outside of the United States. In addition, studies thus far have examined the effectiveness of honey as a wound treatment and have failed to evaluate patient care satisfaction with honey as a treatment option and the treatment costs associated with the use of honey in clinical care. These two outcomes can provide valuable insight into the appropriateness and feasibility of using honey in everyday clinical care. Overall, information obtained from this study will yield knowledge on the potential benefits of this product for burn wound treatment compared to standard care (i.e., SANTYL®).

ELIGIBILITY:
Inclusion Criteria:

* New patient presenting with a partial thickness burn injury in at least two non-contiguous locations of the body.
* Enrollment will occur within 72 hours of sustaining a burn injury.

Exclusion Criteria:

* Cognitive or language barriers that preclude completion of study measures.
* Have burn injuries exceeding 40% total body surface area (TBSA).
* Have a diagnosis of immunodeficiency or kidney disease.
* Are receiving treatment (e.g., chemotherapy, dialysis) that can create concerns with immunodeficiency or affect healing.
* Are pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-03-15 (Actual); Primary Completion 2016-08-18 (Actual); Study Completion 2016-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel M Aballay, MD, Principal Investigator — Western Pennsylvania Hospital Burn Center; Christina L Duncan, PhD, Principal Investigator — West Virginia University
Locations (1):
- Western Pennsylvania Hospital Burn Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Molan PC. The evidence and the rationale for the use of honey as a wound dressing. Wound Practice and Research, 19(4): 204-220, 2011.
- [Background] Blair SE, Cokcetin NN, Harry EJ, Carter DA. The unusual antibacterial activity of medical-grade Leptospermum honey: antibacterial spectrum, resistance and transcriptome analysis. Eur J Clin Microbiol Infect Dis. 2009 Oct;28(10):1199-208. doi: 10.1007/s10096-009-0763-z. Epub 2009 Jun 10. PMID 19513768
- [Background] George NM, Cutting KF. Antibacterial Honey (Medihoney): in-vitro Activity Against Clinical Isolates of MRSA, VRE, and Other Multiresistant Gram-negative Organisms Including Pseudomonas aeruginosa. Wounds. 2007 Sep;19(9):231-6. PMID 25942744
- [Background] Cooper RA, Halas E, Molan PC. The efficacy of honey in inhibiting strains of Pseudomonas aeruginosa from infected burns. J Burn Care Rehabil. 2002 Nov-Dec;23(6):366-70. doi: 10.1097/00004630-200211000-00002. PMID 12432313
- [Background] Cooper RA, Jenkins L, Henriques AF, Duggan RS, Burton NF. Absence of bacterial resistance to medical-grade manuka honey. Eur J Clin Microbiol Infect Dis. 2010 Oct;29(10):1237-41. doi: 10.1007/s10096-010-0992-1. Epub 2010 Jun 13. PMID 20549529
- [Background] Gupta SS, Singh O, Bhagel PS, Moses S, Shukla S, Mathur RK. Honey dressing versus silver sulfadiazene dressing for wound healing in burn patients: a retrospective study. J Cutan Aesthet Surg. 2011 Sep;4(3):183-7. doi: 10.4103/0974-2077.91249. PMID 22279383
- [Background] Baghel PS, Shukla S, Mathur RK, Randa R. A comparative study to evaluate the effect of honey dressing and silver sulfadiazene dressing on wound healing in burn patients. Indian J Plast Surg. 2009 Jul;42(2):176-81. doi: 10.4103/0970-0358.59276. PMID 20368852
- [Background] Malik KI, Malik MA, Aslam A. Honey compared with silver sulphadiazine in the treatment of superficial partial-thickness burns. Int Wound J. 2010 Oct;7(5):413-7. doi: 10.1111/j.1742-481X.2010.00717.x. PMID 20649832

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited largely from an outpatient burn care clinic in a hospital in the Northeastern U.S.. Some participants also were recruited during their hospitalization in the hospital's inpatient burn care center. The first participant was enrolled on 03/15/2014; the final participant was enrolled on 08/11/2016.
Groups:
- Medihoney & Santyl: Each patient received both interventions simultaneously, but on non-contiguous parts of the body (e.g., bilateral lower extremities), each with partial thickness burns of similar depth. One intervention was MEDIHONEY® GEL WITH ACTIVE LEPTOSPERMUM HONEY, a moist dressing made of Active Leptospermum Honey (+15) in combination with natural gelling agents. MEDIHONEY® GEL dressings contains 80% honey. The other intervention was SANTYL®, an FDA-approved sterile enzymatic debriding ointment which contains 250 collagenase units per gram of white petrolatum USP.
Period: Overall Study
Arm/Group | Medihoney & Santyl
Started | 21
Completed | 13
Not Completed | 8
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 5
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Total enrolled = 21. Only one pediatric participant was enrolled in this study. As an outlier, this participant was removed from all analyses. Another participant had missing data for all baseline measurement. Thus, total analyzed at baseline = 19.
Groups:
- Medihoney & Santyl: Each patient received both interventions simultaneously, but on non-contiguous parts of the body (e.g., arm vs. leg), each with partial thickness burns of similar depth. One intervention was MEDIHONEY® GEL WITH ACTIVE LEPTOSPERMUM HONEY, a moist dressing made of Active Leptospermum Honey (+15) in combination with natural gelling agents. MEDIHONEY® GEL dressings contains 80% honey. The dressing has a low pH and can help to lower the overall pH of wounds. The dressing also possesses a high osmotic potential, which assists in debridement. The other intervention was SANTYL®, an FDA-approved sterile enzymatic debriding ointment which contains 250 collagenase units per gram of white petrolatum USP. SANTYL® Ointment is indicated for debriding chronic dermal ulcers and severely burned areas.
Arm/Group | Medihoney & Santyl
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Total enrolled = 21. Only one pediatric participant was enrolled in this study. As an outlier, this participant was removed from all analyses. Another participant had missing data for all baseline measurement. Thus, total analyzed at baseline = 19.
  years | 42.00 (14.24)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Total enrolled = 21. Only one pediatric participant was enrolled in this study. As an outlier, this participant was removed from all analyses. Another participant had missing data for all baseline measurement. Thus, total analyzed at baseline = 19.
  Participants
    Female | 7
    Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Total enrolled = 21. Only one pediatric participant was enrolled in this study. As an outlier, this participant was removed from all analyses. Another participant had missing data for all baseline measurement. Thus, total analyzed at baseline = 19.
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 10
    Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Total enrolled = 21. Only one pediatric participant was enrolled in this study. As an outlier, this participant was removed from all analyses. Another participant had missing data for all baseline measurement. Thus, total analyzed at baseline = 19.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 3
    White | 16
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Population: Total enrolled = 21. Only one pediatric participant was enrolled in this study. As an outlier, this participant was removed from all analyses. Another participant had missing data for all baseline measurement. Thus, total analyzed at baseline = 19.
  participants
    United States | 19
Cause of Burn Injury [Count of Participants; unit: Participants] — Classification for cause of burn injury; measured by medical chart review Population: Total enrolled = 21. Only one pediatric participant was enrolled in this study. As an outlier, this participant was removed from all analyses. Another participant had missing data for all baseline measurement. Thus, total analyzed at baseline = 19.
  Participants
    Thermal | 10
    Scald | 5
    Contact | 4
Total Body Surface Area Burned [Mean (Standard Deviation); unit: Total body surface area percentage] — Measured via medical chart review Population: Total enrolled = 21. Only one pediatric participant was enrolled in this study. As an outlier, this participant was removed from all analyses. Another participant had missing data for all baseline measurement. Thus, total analyzed at baseline = 19.
  Total body surface area percentage | 4.75 (4.57)

OUTCOME MEASURES:

1. Primary Outcome: Change in Wound Appearance
Description: Pictures of wounds and associated "seepage test" paper towels, without indication of date or arm of treatment, were rated by two independent physicians regarding healed or not yet healed. This information was then be used to calculate a "time to heal" variable (# of days) for each patient.
Time Frame: Daily for 7 to 21 days, depending on time it takes burn injury to completely heal
Population: Each participant received both arms of treatment to control for individual healing factors (thus, this is a single group study). Initial analyses yielded inconclusive agreement on healing time due to low quality of pictures (e.g., lighting, focus) and physician reported difficulty in using still photos in isolation to judge wound healing.
Groups:
- Medihoney & Santyl: Each patient received both interventions (MEDIHONEY® GEL & SANTYL® Ointment) simultaneously, but on non-contiguous parts of the body that each consisted of partial thickness burn injuries of similar depth. For example, if a patient presented with bilateral second-degree burns to the lower extremities, one leg was treated with MEDIHONEY® GEL with Active leptospermum honey dressing, while the other leg was treated with SANTYL® ointment dressing.
Arm/Group | Medihoney & Santyl
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Presence vs. Absence of Bacteria in Burn Wound
Description: Wound swab culture results will be compared between treatment modalities via a McNemar test, with treatment modality (MEDIHONEY® GEL versus SANTYL® ointment) and outcome (Positive versus Negative wound culture results for presence of Pseudomonas aeruginosa and/or other bacteria) as the independent and dependent variables, respectively. Each participant has two wound cultures, one for MEDIHONEY® GEL and one for SANTYL® ointment.
Time Frame: Day 7 of study
Population: Each participant received both arms of treatment to control for individual healing factors (thus, this is a single group study & McNemar test is used). Seven participants had missing wound culture data for one or both treatment conditions.
Measure: Number; unit: participants
Groups:
- MEDIHONEY: Each patient received both interventions (MEDIHONEY® GEL & SANTYL® Ointment) simultaneously, but on non-contiguous parts of the body that each consisted of partial thickness burn injuries of similar depth. For example, if a patient presented with bilateral second-degree burns to the lower extremities, one leg was treated with MEDIHONEY® GEL with Active leptospermum honey dressing, while the other leg was treated with SANTYL® ointment dressing. This arm will be MEDIHONEY ® GEL.
- SANTYL: Each patient received both interventions (MEDIHONEY® GEL & SANTYL® Ointment) simultaneously, but on non-contiguous parts of the body that each consisted of partial thickness burn injuries of similar depth. For example, if a patient presented with bilateral second-degree burns to the lower extremities, one leg was treated with MEDIHONEY® GEL with Active leptospermum honey dressing, while the other leg was treated with SANTYL® ointment dressing. This arm will be SANTYL ® Ointment.
Arm/Group | MEDIHONEY | SANTYL
Number analyzed (Participants) | 13 | 13
participants
  Negative Wound Culture | 1 | 1
  Positive Wound Culture | 12 | 12
Statistical Analysis 1: Comparison: MEDIHONEY; Each participant received both treatment modalities - MEDIHONEY® and SANTYL - and thus had two wound cultures performed, one for each treatment modality. This was a single group study; however, wound culture results were contrasted with each other across participants. Thus, independent variable was treatment modality, while dependent variable was the wound culture result (positive for presence of bacteria versus negative for absence of bacteria); Test type: Superiority; p = 1.00, McNemar — A priori threshold for statistical significance was p<0.05. Each case (participant) serves as its own control because they received both treatment modalities simultaneously; McNemar test was used because participants received both treatments, so this variable was non-independent in our single group sample; Odds Ratio (OR) = 1.000 — 2-sided

3. Other Pre Specified Outcome: Patient Satisfaction Questionnaire Score at End of Study Participation
Description: Patients rated their experience separately for MEDIHONEY & SANTYL treatment. Responses were 6-point Likert type ratings across 6 items measuring pain, burn appearance, ease of use, and willingness to recommend that treatment to other patients. Potential score range was 6-36, with higher scores representing greater satisfaction.The mean difference in participant satisfaction for the MEDIHONEY® GEL and SANTYL® ointment treatments was assessed via a within-subject, two-tailed t-test.
Time Frame: 7 to 21 days after enrollment, depending on time it takes for burn injury to completely heal or to discontinue study participation
Population: Each participant received both treatment arms (single group study). To reduce bias in results, participants not lost to follow-up were asked to complete this survey, regardless of whether they completed the study or discontinued participation due to withdrawal, need for treatment change, or adverse event. Six participants were missing this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medihoney & Santyl
Number analyzed (Participants) | 14
score on a scale
  MEDIHONEY | 30.86 (2.07)
  SANTYL | 28.00 (3.16)
Statistical Analysis 1: Comparison: Medihoney & Santyl; A paired samples, 2-tailed, t-test was used to compare means within participants for ratings of MEDIHONEY and SANTYL satisfaction total scores. The null hypothesis was that the two mean scores would not differ significantly at p<.05 level; Test type: Superiority; p = .003, t-test, 2 sided — The null hypothesis was that the two mean scores would not differ significantly at p<.05 level; df = 13; Mean Difference (Final Values) = 3.615, 95% CI 2-sided [1.149 to 4.565], Standard Error of Mean .790

4. Other Pre Specified Outcome: Cost of Treatment (MEDIHONEY vs. SANTYL) Supplies
Description: The total treatment costs for MEDIHONEY® GEL and SANTYL® ointment will be summed across participants. The total number of SANTYL® tubes and MEDIHONEY® GEL patches used will be totaled for each participant, multiplied by cost, and then compared within subjects with a paired samples, t-test.
Time Frame: At the end of treatment, which can last from 7 to 21 days after enrollment
Population: We did not analyze these data because we determined later that the values were confounded by multiple uncontrolled factors - i.e., size of the burn, unstandardized patient variation in amount of cream used (as treatment was performed at home). Normalizing values to burn size would not be sufficient to make valid comparison.
Arm/Group | Medihoney & Santyl
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of enrollment until the time of study completion, i.e., when wounds were healed, or study discontinuation due to participant withdrawing from research or experiencing an adverse event. Given expected healing time for these depth of burn wounds, adverse event data were gathered for up to 4 weeks after enrollment across all participants.
Description: Data were collected via physician examination during weekly follow-up clinic or hospital visits at days 7, 14, or 21 or during an unscheduled follow-up clinic visit (for outpatients) prompted by patient concerns (e.g., calling clinic to express concern about wound appearance). Adverse events were recorded in a log and reported to the IRB, per institutional standards.
Groups:
- Medihoney: MEDIHONEY® was the target treatment for this arm. However, each patient received both interventions (MEDIHONEY® GEL & SANTYL® Ointment) simultaneously, but on non-contiguous parts of the body that each consisted of partial thickness burn injuries of similar depth, to control for individual healing factors when comparing the treatments. For example, if a patient presented with bilateral second-degree burns to the lower extremities, one leg was treated with MEDIHONEY® GEL with Active leptospermum honey dressing, while the other leg was treated with SANTYL® ointment dressing.
- Santyl: SANTYL® was the target treatment for this arm However, each patient received both interventions (MEDIHONEY® GEL & SANTYL® Ointment) simultaneously, but on non-contiguous parts of the body that each consisted of partial thickness burn injuries of similar depth, to control for individual healing factors when comparing the treatments. For example, if a patient presented with bilateral second-degree burns to the lower extremities, one leg was treated with MEDIHONEY® GEL with Active leptospermum honey dressing, while the other leg was treated with SANTYL® ointment dressing.
Arm/Group | Medihoney | Santyl
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medihoney (N=21) | Santyl (N=21)
Infection of the burn wound precipitating change in treatment to include prescribed antibiotics (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Positive wound cultures do not necessarily indicate adverse event (AE) because of normal expected flora. Thus, AE was defined as only infections developing in the burn wound that precipiated a change in treatment to include prescribed antibiotics.

LIMITATIONS AND CAVEATS:
Early termination resulting from strict inclusion criteria reduced sample size for analysis; Technical & methodological problems in measurement (photos to gauge healing; treatment costs confounded by variation in gel use) led to uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes